CLINICAL TRIAL: NCT06192966
Title: Efficacy of a Food Supplement for the Treament of Recurrent Urinary Tract Infections
Brief Title: Effect of Probiotics on Recurrent Urinary Tract Infections
Acronym: CYSCARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participants meeting selection criteria
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AB-CYSCARE
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Urinary Tract Infections
Keywords: Probiotics; Women health; Microbiota
MeSH Terms: conditions — Urinary Tract Infections | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Probiotic and placebo products will be provided in identical packaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Probiotic formulation comprising Lactobacillus plantarum CECT8675 and CECT8677 in combination with cranberry, and vitamine C in a capsule format. Probiotic strains have Qualified Presumption of Safety (QPS) sttus by European Food Safety Authority.
  Interventions: Dietary Supplement: Food supplement
- Placebo (Placebo Comparator): Placebo composed of maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Food supplement — Probiotic formulation containing Lactobacillus plantarum, cranberry and vitamine C for 6 months 1 capsule/day
  Arms: Experimental
Dietary Supplement: Placebo — Placebo composed of maltodextrin for 6 months 1 capsule/day
  Arms: Placebo

SUMMARY:
Randomized clinical trial to evaluate the effect of a probiotic mixture of Lactobacillus plantarum on recurrent urinary tract infections in women. Secondary outcomes comprise variation in vaginal/perianal microbiota, product tolerability, safety and consumer's satisfaction with the product.

DETAILED DESCRIPTION:
Double-blind, randomized, placebo-controlled clinical trial to determine the effect of two probiotic strains of Lactobacillus plantarum on recurrent urinary tract infections in women. Women are randomized 1:1 to one of the following study groups: one group will receive a capsule/day of the mixture of Lactobacillus plantarum in combination with cranberry, and vitamine C; and the other group will receive a capsule of placebo for 6 months. Main study outcome is the number of women who have recurrence of UTIs during th estudy compared to the placebo group. Secondary outcomes comprise the duration of disease free period, duration and severity of symptomatology, the number of symptomatic UTIs during the study, variation of Lactobacillus plantarum levels in the vaginal/perianal microbiota, product tolerability, safety and consumer's satisfaction with the product.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age.
* Women who have had at least one episode of UTI in the past 4 months
* Women with a well-documented history of recurrent UTIs: ≥2 infections in the past 6 months or ≥3 in the past 12 months.
* Women who have been treated with an antibiotic regimen for each episde of UTI
* Recurrence due to reinfection, not relapse: multiple infections should be spaced by a minimum of 2 weeks or in case of a shorter time, with negative urine culture between them
* Women who use contraception to prevent pregnancy and who do not plan a pregnancy during the study period

Exclusion Criteria:

* Pregnant or breastfeeding women
* Underlying chronic disease: diabetes mellitus, kidney failure, cancer, spinal cord injury, polycystic ovary
* Women wih catheters in the urethra
* Women who consume probiotics or foods, beverages or supplements containing extracts or parts of the genus Vaccinum sp, including other forms of V. macrocarpon (blueberry), V. myrtillus (European blueberry), V. angustifolium (wild or low buch blueberry), V. corymbosum (tall bch blueberry) or V. vitis-ideae (mountain blueberry) during the 2 weels prior to recruitment.
* High consumption of fruits rich in phenolic compounds, with special reference, to berries
* Women allergic to red fruits

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 106 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Recurrence of Urninary Tract Infections (UTIs) | month 6
  Number of women who have recurrence of UTIs

SECONDARY OUTCOMES:
Time without UTI | month 6
  Time (in days) disease free until the next UTI
Total symptomatic UTIs number | month 6
  Number of symptomatic UTIs
Change in UTI symptomatology | baseline, month 6
  Change in the presence of UTI-related list of symptoms documented in CRF as "yes" or "no"
Change in Microbiota | baseline, month 6
  Change in Lactobacillus plantarum levels in the vaginal/perianal microbiota
Incidence of Treatment-Emergent Adverse Events | From baseline until month 6
  Assessed by the reporting of Adverse Events
Satisfaction with the product | Month 6
  Consumer's satisfaction with the product assessed through Likert scale (ranging from very unsatisfied to very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Prieto González, MD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (4):
- Spain (4):
  - Fundació Puigvert, Barcelona, Barcelona
  - Hospital Universitario de Caceres, Cáceres, Cáceres
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario Virgen de Arrixaca, Murcia, Murcia

IPD SHARING:
Plan to Share IPD: No